CLINICAL TRIAL: NCT07233304
Title: Incidence of Complications From the Alveolar Opening Maneuver in Mechanically Ventilated Children With Respiratory Distress Syndrome
Brief Title: Complications of the Alveolar Opening Maneuver in Children on Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: Hospital de Alta Complejidad en Red (Other)
Responsible Party: Principal Investigator, Belen Castelli, Physical Therapy, Hospital de Alta Complejidad en Red
Other Study IDs: 080-2025-EO
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Positive End-expiratory Pressure (PEEP); Oxygenation Index; Pediatric Intensive Care Unit; Pediatric Acute Lung Injury; Respiratory Distress Syndrome, Pediatric; Complication
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alveolar Opening Maneuver and PEEP Titration (AOM+P): Patients under invasive mechanical ventilation for pediatric acute respiratory distress syndrome (PARDS) who undergo a standardized alveolar opening maneuver followed by decremental PEEP titration according to institutional protocol. The maneuver consists of stepwise increases in PEEP until reaching a plateau pressure of 35 cmH₂O (or up to 40 cmH₂O in patients with reduced chest wall compliance), maintained for 2 minutes, followed by decremental PEEP titration to determine the optimal level based on driving pressure and oxygen saturation. The procedure is performed once clinically indicated, with continuous hemodynamic and oxygenation monitoring.
  Interventions: Procedure: Alveolar Opening Maneuver and PEEP Titration (AOM+P)

INTERVENTIONS:
Procedure: Alveolar Opening Maneuver and PEEP Titration (AOM+P) — Standardized ventilatory procedure performed in pediatric patients under invasive mechanical ventilation with acute respiratory distress syndrome (PARDS). The intervention consists of a controlled alveolar opening maneuver with stepwise PEEP increments up to a plateau pressure of 35 cmH₂O (or up to 40 cmH₂O in patients with reduced chest wall compliance), maintained for 2 minutes, followed by a decremental PEEP titration to determine the optimal PEEP level based on driving pressure and oxygenation response. The procedure is performed once clinically indicated, under continuous hemodynamic and oxygen monitoring, according to the institutional safety protocol.
  Other Names: Alveolar Opening Protocol, PEEP Titration Procedure, AOM+P Institutional Protocol

SUMMARY:
The objective of this research is to analyze the overall incidence of complications associated with a therapeutic maneuver known as alveolar opening and subsequent titration of positive end-expiratory pressure (PEEP) in pediatric patients with acute respiratory distress syndrome (ARDS). These procedures are part of the standard care provided in the Pediatric Intensive Care Unit (PICU) and are used to improve pulmonary oxygenation and respiratory mechanics. Through this study, we aim to gather information that will help improve the safety and effectiveness of these interventions in critically ill patients.

DETAILED DESCRIPTION:
Objective

To analyze the overall incidence of complications associated with alveolar opening maneuvers and PEEP in pediatric patients with respiratory distress syndrome.

Materials and Methods

Study setting A prospective cohort study will be conducted between April and September in the Pediatric Intensive Care Unit (PICU) of the Hospital Cuenca Alta Néstor Kirchner (HCANK).

Sample All patients meeting the eligibility criteria will be included. An estimated total of 143 maneuvers involving alveolar opening maneuversand PEEP are to be analyzed, as these procedures are part of the standard care in managing ventilated patients with ARDS and are included in the institutional protocol (see Appendix).

Inclusion criteria:

* Patients under 14 years of age admitted to the HCANK PICU
* More than 4 hours of invasive mechanical ventilation (IMV)
* An oxygenation index (OI) ≥4 or an oxygen saturation index (OSI) ≥5
* Indication for alveolar opening maneuvers and PEEP as determined by the treating team

Exclusion criteria:

* Predicted body weight (PBW) >45.5 kg
* Recent pulmonary resection surgery (<7 days)
* Presence of broncho-pleural fistula or peri-tube leak >25% of the tidal volume
* Hemoglobin decline <7 g/dL
* Patients with congenital or acquired heart diseases with significant intracardiac shunt

Variables:

Outcome variable:

- Overall incidence of complications related to alveolar opening maneuvers and PEEP

Procedure Once patients are included, demographic, clinical, and relevant background data will be recorded in a dedicated data sheet. Following this, study evaluators will record baseline clinical data from the multiparameter monitor prior to performing the alveolar opening maneuvers and PEEP procedures. Relevant values will be obtained from the advanced monitoring sheet completed by the treating team.

During the alveolar opening maneuvers and PEEP procedures, intra-procedural complications will be noted, and monitoring will continue for 4 hours after the procedure to observe for any complications that develop.

If, due to intercurrences or the treating team's decision, the alveolar opening maneuvers and PEEP need to be repeated before 4 hours, monitoring will still continue for 4 hours after the last maneuver.

Statistical Analysis Categorical variables will be described using absolute numbers and percentages of the total, while continuous variables will be expressed using measures of central tendency and dispersion or position, depending on their distribution.

The Kolmogorov-Smirnov test will be used as a goodness-of-fit test to determine the distribution of numerical variables.

To address the objective, the overall incidence of complications will be calculated, with estimates and 95% confidence intervals provided.

Data analysis will be performed using IBM SPSS Windows version 25.0 (IBM Corp., Armonk, NY, USA), R version 3.6.3 (R Core Team, 2020), and the ggplot2 package version 3.3.2 (Wickham, 2016) for graph creation.

Sample size calculation The calculation assumes a null hypothesis where the incidence of complications after alveolar opening maneuvers and PEEP is 5%, based on previously reported data indicating a lower rate of complications.

The alternative hypothesis posits that the incidence of complications related to alveolar opening maneuvers and PEEP is less than 5%.

A total of 143 maneuvers are planned to be recruited according to the sample size calculation based on these hypothesized values.

ELIGIBILITY:
Inclusion criteria:

* Patients under 14 years of age admitted to the HCANK PICU
* More than 4 hours of invasive mechanical ventilation (IMV)
* An oxygenation index (OI) ≥4 or an oxygen saturation index (OSI) ≥5
* Indication for ARM and PEEP as determined by the treating team

Exclusion criteria:

* Predicted body weight (PBW) >45.5 kg
* Recent pulmonary resection surgery (<7 days)
* Presence of broncho-pleural fistula or peri-tube leak >25% of the tidal volume
* Hemoglobin decline <7 g/dL
* Patients with congenital or acquired heart diseases with significant intracardiac shunt.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients under 14 years of age admitted to the Pediatric Intensive Care Unit (PICU) of the Hospital Cuenca Alta Néstor Kirchner
Sampling Method: Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of complications related to the alveolar opening maneuver and PEEP titration | 4 hours post-procedure
  The number and proportion of patients who develop any adverse event directly associated with the alveolar opening maneuver or PEEP titration within 4 hours after the procedure. Complications may include hemodynamic instability (e.g., hypotension, bradycardia), oxygen desaturation, barotrauma (such as pneumothorax), or cardiac arrhythmias observed during or after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Garcia Urrutia, BCS, Principal Investigator — Hospital de Alta Complejidad Cuenca Alta "Néstor Kirchner", Buenos Aires, Argentina; Belen Castelli, BCS, Principal Investigator — Hospital de Alta Complejidad Cuenca Alta "Néstor Kirchner", Buenos Aires, Argentina
Locations (1):
- Hospital Cuenca Alta Néstor Kirchner, Cañuelas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No